CLINICAL TRIAL: NCT01790906
Title: Safety and Effectiveness Study of Percutaneous Catheter-base Renal Sympathetic Denervation for Patients With Chronic Heart Failure
Brief Title: Renal Sympathetic Denervation for Patients With Chronic Heart Failure
Acronym: RSD4CHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qijun Shan, Professor,Director, Cardiac Arrhythmia Group, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-SR-001
Record Dates: First submitted 2013-02-07; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Renal Sympathetic Denervation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSD+Conventional therapy (Active Comparator): We will recruit 100 randomised CHF patients who meet the inclusion criteria.First undergo renal artery angiography procedure to confirm anatomy.If renal artery meet the inclusion criteria,give the renal sympathetic denervation.At the same time, we will use conventional therapy to protect cardiac function.then we will conduct a clinic follow-up and a telephone follow-up.
  Interventions: Procedure: RSD; Other: Conventional therapy
- Conventional therapy (Placebo Comparator): We also will recruit 100 randomised CHF patients who meet the inclusion criteria.there are no significant differences in age,gender,race,past medical history,personal history and so on between the two groups.In this group we will use therapy just like the RSD+Conventional therapy group.we will conduct a clinic and a telephone follow-up.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Procedure: RSD — Contrast renal angiography was performed to localize and assess the renal arteries for accessibility and appropriateness for RSD .once the anatomy was deemed acceptable, the internally irrigated radiofrequency ablation catheter(Celsius Thermocool,Biosense Webster,Diamond Bar,California)was introduced into each renal artery.then was maneuvered within the renal artery to allow energy delivery in a circumferential,longitudinally staggered manner to minimize the chance of renal artery stenosis.About six to nine ablation at 10W for 1 min each were performed in both renal arteries.during ablation, the catheter system monitored tip temperature and impedance,altering radiofrequency energy delivery in response to predetermined algorithm.
  Other Names: renal sympathetic denervation; renal denervation; renal ablation
  Arms: RSD+Conventional therapy
Other: Conventional therapy — Optimizing drug therapy,included angiotensin-converting enzyme inhibitors,aldosterone antagonist,beta-receptor blockers,diuretic,digoxin and so on.The patients with chronic heart failure ,whos'condition need for CRT-D(cardiac resynchronization therapy )/ICD(implantable cardioverter-defibrillator),are considered to implant CRT/ICD .CRT is abbreviation for cardiac resynchronization therapy ,ICD is defined for Implantable Cardioverter defibrillator.

SUMMARY:
To study whether renal sympathetic denervation(RSD) RSD can slow the progression of CHF and reduce the rate of all-cause mortality effectively and securely.

DETAILED DESCRIPTION:
Chronic heart failure(CHF) as the final stage of various heart diseases is a global and growing public health problem, and its morbidity increases with age. At present, the main therapies for CHF contain drug therapy (including angiotensin-converting enzyme inhibitors, aldosterone antagonist, beta-receptor blockers, diuretic, digoxin etc ) , CRT-D(cardiac resynchronization therapy )/ICD(implantable cardioverter-defibrillator), biological treatment, ultrafiltration dialysis, heart transplantation and so on. Optimize drug therapy is the foundation of CHF, but hypotension and bradycardia limit its indications. ESC(European Society of Cardiology)/AHA(American Heart Association) guidelines recommended CRT-P/D and ICD for drug resistant CHF, but the financial burden limit the use of them and some patients have no response to them. Donors and high costs are considered as two problems which limit heart transplantation appeal. Above all, we are always searching for a new treatment strategy for patients with chronic heart failure. Chronic over-activation of sympathetic nervous system is a major component of heart failure and involves efferent and afferent pathways between brain and many organs. Recently, some studies in animals and humans suggest that activation of both efferent and afferent renal nerves play a crucial role in the pathogenesis and progression of CHF. Activation of renal nerves in CHF may cause a reflex increase in sympathetic tone that contributes to elevated peripheral vascular resistance and vascular remodeling as well as left ventricular remodeling and dysfunction. Recently, many clinical trials have corroborated that catheter-based renal sympathetic denervation (RSD) significantly decreased sympathetic-nerve activity (MSNA) in muscle and whole-body, with a decrease in renal and whole-body norepinephrine spillover. Simultaneously, many clinical researches have also verified that RSD can safely be used to control hypertension, reduce left ventricular hypertrophy, improve glucose tolerance impaired ,decrease proteinuria and sleep apnea severity, which are all recognized as independent risk factors for the development and progression of CHF. Therefore, this randomized parallel control clinical trial was designed to demonstrate whether RSD can slow the progression of CHF and reduce the rate of all-cause mortality effectively and securely.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is ≥18 and ≤ 75 years of age
2. Individual has a history of heart failure more than half a year
3. Individual's Cardiac function is betweenⅡ-Ⅳlevel(NYHA)
4. Ejection fraction ≦ 35%
5. Renal artery CTA (computed tomographic arteriography)inspection renal artery length ≧ 2 cm, diameter ≧ 4 mm, no single double renal artery, renal artery start without distortion/tumor sample expansion,ect
6. Individual agrees to have all study procedures performed and is competent and willing to provide written,informed consent to participate in this clinical study

Exclusion Criteria:

1. Individual has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.
2. Individual has experienced renal artery stenosis,or A history of prior renal artery intervention including balloon angioplasty or stenting.
3. Individual has an estimated glomerular filtration rate (eGFR) of < 45mL/min/1.73m2, using the MDRD(Modification of Diet in Renal Disease) calculation.
4. Individual has Acute heart failure.
5. Individual has experienced a cerebrovascular accident within 3 months of the screening visit, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
6. Individual has experienced sick sinus syndrome.
7. Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia, or arrhythmias such as atrial fibrillation).
8. Individual is pregnant, nursing or planning to be pregnant. [Female participants of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to treatment.]
9. Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
10. Individual is currently enrolled in another investigational drug or device trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality,Cardiovascular events | 24 months
  To study effect of renal sympathetic denervation(RSD)on All-cause mortality ad cardiovascular events(cardiac death ,myocardial infarction ,malignant arrhythmia,angina and so on)

SECONDARY OUTCOMES:
Blood pressure | 24 months
  To study the effect of renal sympathetic denervation on blood pressure in patients with hypertension,which can be measured by ambulatory blood pressure and home pressure monitoring.
Life quality and symptom | 24 months
  Life quality on 36-item short-form(SF-36)will be carried out during the follow-up to study the patients' life quality.Symptom will also be carried out by six walk distance during the follow-up,
Rehospitalization rate | 24 months
  To study whether RSD can reduce the patients'rehospitalization rate because of heart failure,which will be measured by questionnaire and telephone follow-ups.
The recurrence rate of electric storm with ICD | 24 months
  To study the recurrence rate of electric storm with ICD ,which will be measured by questionnaire and telephone follow-ups.
Cardiac function an structure | 24 months
  The effect of renal sympathetic denervation(RSD)on cardiac function and structure can be measured by the six-minute walking test and echocardiographic(include left ventricular ejection fraction,left ventricular end diastolic diameter,ventricular septal thickness ), NYHA functional class,BNP(brain-type natriuretic peptide).

CONTACTS AND LOCATIONS:
Overall Officials: Shan Qijun, Professor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Meddical University, Nanjing, Jiangsu, China